CLINICAL TRIAL: NCT06102239
Title: New Diagnostic Markers In Dignosis Of Complicated Appendix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Mohamed Amin, Residiant in general surgery department, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Soh-Med-23-09-08Ms
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Complicated Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Bilirubin level sodium level c reactive protein level — detect level of bilirubin,sodium &c-reactive protein as indicator of complicated appendicitis

SUMMARY:
Most common cause of acute abdomen is acute appendicitis delay dignosis of acute appendicitis lead to complications as perforation this study examined efficacy of hyperbilirubinemia&hyponatremia as indicator of complicated appendicitis

ELIGIBILITY:
Inclusion Criteria:

* all patient admitted for acute appendicitis underwent surgery and post operativly confirmed histopathology of acute appendicitis

Exclusion Criteria:

* patient with liver disease Liver transplantation Chronic alcoholism Congental biliary disease Pregnancy Appendicular neoplasm Hemolytic disease Hepatocellular carcinoma

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Level of bilirubin in acute appendicitis | 6 months
Level of sodium in acute appendicitis | 6 months
Level of c-reactive proteins in acute appendicitis | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Virmani S, Prabhu PS, Sundeep PT, Kumar V. Role of laboratory markers in predicting severity of acute appendicitis. Afr J Paediatr Surg. 2018 Jan-Mar;15(1):1-4. doi: 10.4103/ajps.AJPS_47_16. PMID 30829300
- [Background] Kar S, Behera TK, Jena K, Sahoo AK. Hyperbilirubinemia as a Possible Predictor of Appendiceal Perforation in Acute Appendicitis: A Prospective Study. Cureus. 2022 Feb 2;14(2):e21851. doi: 10.7759/cureus.21851. eCollection 2022 Feb. PMID 35282512
- [Background] Alvarado A. A practical score for the early diagnosis of acute appendicitis. Ann Emerg Med. 1986 May;15(5):557-64. doi: 10.1016/s0196-0644(86)80993-3. PMID 3963537
- [Background] Kanumba ES, Mabula JB, Rambau P, Chalya PL. Modified Alvarado Scoring System as a diagnostic tool for acute appendicitis at Bugando Medical Centre, Mwanza, Tanzania. BMC Surg. 2011 Feb 17;11:4. doi: 10.1186/1471-2482-11-4. PMID 21329493